CLINICAL TRIAL: NCT03620058
Title: Phase 1 Study of Autologous Anti-CD22 Chimeric Antigen Receptor Redirected T Cells (CART22-65s) Alone and When Co-administered With Humanized Anti-CD19 Chimeric Antigen Receptor Redirected T Cells (huCART19) In Patients With Chemotherapy Resistant Or Refractory Acute Lymphoblastic Leukemia
Brief Title: CART22 Alone or in Combination With huCART19 for ALL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 830049; UPCC #12418
Record Dates: First submitted 2018-06-25; First posted 2018-08-08 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Chemotherapy Resistant Acute Lymphoblastic Leukemia; Refractory Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CART22-65s monotherapy (Experimental)
  Interventions: Biological: CART22-65s cells
- CART22-65s in combination with huCART19 (Experimental)
  Interventions: Biological: CART22-65s cells; Biological: huCART19 Cells

INTERVENTIONS:
Biological: CART22-65s cells — Autologous T cells transduced with a lentiviral vector to express anti-CD22 scFv TCRz:41BB
Biological: huCART19 Cells — Autologous T cells transduced with lentiviral vector to express anti-CD19 scFv TCRζ:4-1BB
  Arms: CART22-65s in combination with huCART19

SUMMARY:
This is a single center, open-label, phase 1 study to determine the safety and feasibility of infusing CART22-65s with or without huCART19 after administration of lymphodepleting chemotherapy in adult patients with relapsed or refractory B-ALL.

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients with relapsed or refractory B cell ALL:

a. Patients with 2nd or greater relapse or refractory to 1st salvage as defined by: i. Recurrent disease in the bone marrow identified morphologically, by immunohistochemistry or by Flow cytometry.

ii. Patients with extramedullary relapse only (no bone marrow involvement) will be eligible if disease response can be assessed radiographically b. Patients with refractory disease as defined by: i. Failure to achieve remission (<5% bone marrow blasts) after 2 cycles of induction chemotherapy ii. Patients that achieve remission but remain MRD+ after ≥2 cycles of induction chemotherapy.

c. Patients with Ph+ ALL are eligible provided they are intolerant to or have failed tyrosine kinase inhibitor therapy.

d. Patients with prior or current history of CNS3 disease* will be eligible only if CNS disease is responsive to therapy.

i. *CNS disease definitions:

1. CNS1 - no blasts seen on cytocentrifuge (CNS negative);
2. CNS2 - total nucleated cell count <5x106/L, but blasts seen on cytocentrifuge;
3. CNS3 - total nucleated cell count 5x106/L with blasts on cytocentrifuge and/or signs of CNS leukemia (i.e. cranial nerve palsy).

   * 2. For Cohort 1: Documentation of CD22 expression on malignant cells at relapse. For Cohort 2: Documentation of CD22 and/or CD19
   * 3. Adequate vital organ function defined as:

     1. Creatinine ≤ 1.6 mg/dl
     2. ALT/AST ≤ 3x upper limit of normal range
     3. Total or Direct bilirubin ≤ 2.0 mg/dl. If Total bilirubin is ≤2.0, Direct bilirubin does not need to be assessed.
     4. Left Ventricle Ejection Fraction (LVEF) ≥ 40% confirmed by ECHO/MUGA
   * 4. Male or female age ≥ 18 years.
   * 5. ECOG Performance Status that is either 0 or 1.
   * 6. No contraindications for leukapheresis.
   * 7. Subjects of reproductive potential must agree to use acceptable birth control methods.

Exclusion Criteria:

* 1. Active hepatitis B or active hepatitis C.
* 2. HIV Infection.
* 3. Class III/IV cardiovascular disability according to the New York Heart Association Classification.
* 4. Subjects with clinically apparent arrhythmia or arrhythmias who are not stable on medical management within two weeks of eligibility confirmation by physician-investigator.
* 5. Active acute or chronic graft-versus-host disease (GVHD) requiring systemic therapy.
* 6. Planned concurrent treatment with systemic steroids or immunosuppressant medications. Patients may be on a stable low dose of steroids (<10mg equivalent of prednisone) for chronic respiratory conditions or adrenal insufficiency. For additional details regarding use of steroid and immunosuppressant medications.
* 7. CNS3 disease that is progressive on therapy, or with CNS parenchymal lesions that might increase the risk of CNS toxicity.
* 8. Pregnant or nursing (lactating) women.
* 10. Patients with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2036-01 (Estimated); Study Completion 2036-01 (Estimated)

PRIMARY OUTCOMES:
Assess the safety of CART22-65s in ALL subjects using the common terminology criteria of adverse events (CTCAE) v5.0. | 15 months
  Frequency and severity of adverse events, including, but not limited to, cytokine release syndrome (CRS).
Assess the safety of combination CART22-65s and huCART19 in relapsed/refractory ALL Subjects using the common terminology criteria of adverse events (CTCAE) v5.0. | 15 months
  Frequency and severity of adverse events, including, but not limited to, cytokine release syndrome (CRS).

SECONDARY OUTCOMES:
Tumor response. | 28 Days
  Overall Complete Remission Rate (ORR) at Day 28 which includes CR and CR with incomplete blood count recovery (CRi).
Tumor response. | 6 months
  overall response rate (CR/CRi by or at Month 6) and disease response status at Month 6
Tumor response. | 1 Year
  overall survival (OS)
Tumor response. | 1 Year
  duration of remission (DOR)
Tumor response. | 1 Year
  relapse free survival (RFS)
Tumor response. | 1 Year
  event free survival (EFS)
CAR T cell kinetics | 1 Year
  Engraftment and persistence in blood by qPCR (or flow cytometry)
CAR T cell kinetics | 1 Year
  Trafficking to target tissue (bone marrow) or other tissues (cerebral spinal fluid and other tissues if available) as determined by qPCR (or flow cytometry).
Evaluate bioactivity of CAR T cells | 1 Year
  Measure levels of systemic soluble immune and inflammatory factors by Luminex-based analyses
Determine antigen expression and normal B cell levels in response to CAR T cells | 1 Year
  Measure CD22, CD19 and B cell levels pre- and post-CAR T cell infusion by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Frey, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Myers RM, DiNofia AM, Li Y, Diorio C, Liu H, Wertheim G, Fraietta JA, Gonzalez V, Plesa G, Siegel DL, Iannone E, Shinehouse L, Brogdon JL, Taylor C, Jadlowsky JK, Hexner EO, Engels B, Baniewicz D, Callahan C, Ruella M, Aplenc R, Barz Leahy A, McClory SE, Rheingold SR, Wray L, June CH, Maude SL, Frey NV, Grupp SA. CD22-targeted chimeric antigen receptor-modified T cells for children and adults with relapse of B-cell acute lymphoblastic leukemia after CD19-directed immunotherapy. J Immunother Cancer. 2025 Apr 17;13(4):e011549. doi: 10.1136/jitc-2025-011549. PMID 40246579